CLINICAL TRIAL: NCT04893421
Title: A Registry Study Evaluating the Magnetic Occult Lesion Localization Instrument (MOLLI) Guidance System for Breast Lesion Localization
Brief Title: Magnetic Occult Lesion Localization Instrument (MOLLI) Guidance System for Breast Lesion Localization
Acronym: MOLLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); North York General Hospital (Other)
Responsible Party: Principal Investigator, Nicole Look Hong, Surgical Oncologist, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 159-2019
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasm
Keywords: Non-palpable lesion; Localization; Lumpectomy; Breast-Conserving Surgery; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: At each site, the first cohort of 25 participants will be treated with the standard of care approach (WGS or RSL) and the subsequent cohort of 25 participants will be treated with MOLLI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care WGS or RSL (No Intervention): Patients will undergo the institutional standard of care approach (WGS or RSL) for BCS. For WGL, a hooked wire will be implanted to mark the center or outer edges of the lesion under imaging guidance. For RSL, patients will be implanted with a radioactive seed using an impregnated needle under imaging guidance. A special handheld probe will be used to find the radioactive seed during the lumpectomy surgery.
- MOLLI Localization (Experimental): Patients will be implanted with a MOLLI seed using a specialized introducer needle under imaging guidance. A special handhold probe and detection system will be used intraoperatively to assist in excision.
  Interventions: Device: MOLLI Localization

INTERVENTIONS:
Device: MOLLI Localization — Patients will be implanted with a MOLLI seed using a specialized introducer needle under imaging guidance. A special handhold probe and detection system will be used intraoperatively to assist in excision.
  Arms: MOLLI Localization

SUMMARY:
The proposed trial is a non-randomized, multi-center, sequential arm registry evaluating clinical, and health economic outcomes following treatment with the Magnetic Occult Lesion Localization Instrument (MOLLI), an approved instrument for Breast Conserving Surgery (BCS) in patients with non-palpable lesions. All patients who have an area of concern in the breast and are identified by their physician as good candidates for BCS are eligible to participate. Patients will eventually be enrolled across 3 surgical sites (Sunnybrook Health Sciences Centre - primary site, Princess Margaret Cancer Centre, and North York General Hospital) over a 2 year period. Patient and system-related outcome measures will first be collected using the centre-specific standard of care (Wire-Guided Localization or Radioactive Seed Localization for BCS) to establish a baseline. Subsequently, centers will transition to the MOLLI system, recording corresponding outcomes to be used for temporal comparison. The overall objective of this study is to evaluate clinical and health economic outcomes with MOLLI compared to standard-of-care approaches.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION

In contemporary breast cancer management, more than 70% of breast cancer patients are eligible for - and select - breast-conserving therapy (BCS). However, issues with cosmesis, patient experience, and treatment workflow efficiency during the therapeutic process have considerable room for improvement.

BCS consists of a surgical procedure whereby the suspicious tumor and a rim of surrounding normal tissue are removed. Up to one-third of all diagnosed breast cancers are non-palpable,and require some form of pre-operative localization to guide precise surgical excision. Currently, options for localization of non-palpable lesions are suboptimal in terms of patient experience, healthcare system resource utilization, and cost-effectiveness.

One of the most common approaches is radioactive seed localization (RSL). RSL consists of insertion of a small radioactive seed under ultrasound guidance to mark the center and/or borders of the tumor. During the procedure the surgeon uses a hand-held probe to detect the seed and guide surgical excision of the lesion intra-operatively. While RSL is effective the use of a radioactive source is and poses many challenges for patients and staff. Another common approach is wired-guided localization (WGL). WGL involves implantation of a hooked wire to mark the center or outer edges of the lesion. Due to modest cost and relative ease of use, WGL use is widespread, however disadvantages include significant patient discomfort, possible migration of the implanted wire, and potential difficulties in localizing axillary lymph nodes.

WHAT ARE THE INVESTIGATORS DOING?

The investigative team of surgeons and scientists are examining an alternative approach to BCS called magnetic occult lesion localization and imaging (MOLLI). Analogous to RSL, this procedure involves implantation of a small passive magnetic seed - under ultrasound or mammographic imaging guidance - directly into or surrounding the tumor; during the procedure the surgeon uses a novel hand-held probe to intra-operatively detect the position of this seed and remove the tumor.

WHY IS THE STUDY BEING CONDUCTED?

MOLLI offers many of the same benefits as RSL but without any radiation. MOLLI also has the potential to be more effective and accurate than other localization methods. MOLLI has recently been evaluated as part of a phase I clinical trial and was demonstrated to be a safe and effective localization technology. The goal for the current trial is to evaluate clinical and health economic outcomes with MOLLI compared to standard-of-care approaches to help improve access to a wireless, low-cost, but effective breast lesion localization technology for breast cancer patients.

WHAT WILL HAPPEN DURING THE STUDY?

As part of this study, researchers will 1) evaluate identify barriers and facilitators related to MOLLI based on feedback from clinical staff, 2) demonstrate cost-effectiveness of MOLLI and 3) gather information on the participants' experience with the MOLLI seed. At each site, the first 25 participants will be treated with the standard of care for BCS (RSL or WGL), and the second 25 participants will be treated with MOLLI.

ARE THERE SIDE EFFECTS?

No side effects are expected from the study treatments. Possible risks associated with using MOLLI include:

A small risk of bleeding A remote risk of allergic reaction to nickel contained in the MOLLI seeds

WHAT WILL HAPPEN AFTER THE STUDY?

Participants may be contacted by a study team member up to and including 16 weeks (6.5 months) after the procedure to take part in a short telephone questionnaire. The questionnaire should take no more than 5 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older with histologically confirmed unifocal breast lesion and identified as a candidate for BCS, this includes patients with high-risk, premalignant (eg. ductal carcinoma in-situ), or malignant (eg. invasive ductal carcinoma) lesions
* Lesions must be non-palpable and require pre-operative localization for surgical guidance
* Lesions must be visible as determined by preoperative breast mammogram and / or ultrasound imaging. Pre-operative MRI is at the discretion of the treating surgeon.

Exclusion Criteria:

* Biologically male patients
* Locally advanced malignant breast cancer
* Any absolute contraindications to BCS
* Pregnancy or lactation
* Existing allergy to metallic seed materials
* Patients requiring MRI after MOLLI seed placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
MOLLI Localization Success Rate | Day 3 (during surgical excision)
  To determine the success rate of localizing the MOLLI seed, along with subsequent accurate removal under MOLLI guidance compared to standard of care approaches.

SECONDARY OUTCOMES:
Specimen Margin Positivity | Day 30
  As reported by anatomical pathology, this metric will evaluate if the excised specimen has negative margins or positive margins.
Re-excision rates | Day 30
  Follow-up will determine if patients required a re-excision / re-operation after determination of positive margin status.
Duration of Excision | Day 3 (during surgery)
  The time required to perform surgical excision of the lesion and MOLLI marker.
Duration of Implantation | Day 1 (localization)
  The duration of MOLLI marker implantation as carried out by the radiologist.
Cost-effectiveness of MOLLI | Day 1 (localization) and Day 3 (post surgery)
  Operating costs and efficiency data of SOC and MOLLI techniques (including disposables, start-up equipment, human resources, timing data for operating and radiology).
Hospital Anxiety and Depression Scale (HADS) to evaluate anxiety and depression | Day 0 (baseline), Day 1 (localization) and Day 30 (1 month follow-up)
  HADS will evaluate anxiety and depression pre and post localization and surgery. Questions will be evaluated on a 4 point scale. Evaluations will occur prior to localization, following localization and approximately 1 month following surgical excision. Higher scores indicate greater anxiety and/or depression.
State-Trait Anxiety Inventory (STAI) to evaluate anxiety | Day 0 (baseline), Day 1 (localization) and Day 30 (1 month follow-up)
  STAI will evaluate anxiety pre and post localization and surgery. Questions will be evaluated on a 4 point scale. Evaluations will occur prior to localization, following localization and approximately 1 month following surgical excision. Higher scores indicate greater anxiety.
Anxiety with Radiation | Day 0 (baseline), Day 1 (localization) and Day 30 (1 month follow-up)
  Anxiety specific to the radioactive seed (for those receiving RSL as the standard of care approach) will be assessed using a questionnaire pre and post localization and surgery. Two questions will be evaluated on a 4 point scale. Evaluations will occur prior to localization, following localization and approximately 1 month following surgical excision. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Look Hong, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Look Hong N, Wright FC, Semple M, Nicolae AM, Ravi A. Results of a phase I, non-randomized study evaluating a Magnetic Occult Lesion Localization Instrument (MOLLI) for excision of non-palpable breast lesions. Breast Cancer Res Treat. 2020 Feb;179(3):671-676. doi: 10.1007/s10549-019-05499-z. Epub 2019 Nov 21. PMID 31754951